CLINICAL TRIAL: NCT01261247
Title: A Phase II Study of the Histone Deacetylase (HDAC) Inhibitor LBH589 (Panobinostat) in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Panobinostat in Treating Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0986; NCI-2010-02326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-004705 (Other: Mayo Clinic IRB); CLBH589BUS59T (Other: Novartis Protocol); MC0986 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Panobinostat; Blotting, Western; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral panobinostat 3 times weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: panobinostat; Other: laboratory biomarker analysis; Genetic: western blotting; Genetic: DNA analysis; Other: flow cytometry; Other: pharmacological study; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: panobinostat — Given orally
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Other: laboratory biomarker analysis — Correlative studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Genetic: DNA analysis — Correlative studies
Other: flow cytometry — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: immunohistochemistry staining method — Optional correlative studies
  Other Names: immunohistochemistry

SUMMARY:
Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well panobinostat works in treating patients with relapsed or refractory non-Hodgkin lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the proportion of confirmed response of LBH589 in patients with relapsed or refractory non-Hodgkin lymphoma. SECONDARY OBJECTIVES: I. To describe the toxicities associated with LBH589 in patients with NHL. II. To evaluate overall survival, progression-free survival, and duration of response in patients treated with LBH589. TERTIARY OBJECTIVES: I. To evaluate the pharmacokinetics of LBH589. II. To assess the correlation between clinical (toxicity and/or tumor response or activity) effects with the pharmacologic (pharmacokinetic/pharmacodynamic) parameters, and/or biologic (correlative laboratory) results. OUTLINE: Patients receive oral panobinostat 3 times weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria

* Biopsy-proven relapsed or refractory non-Hodgkin lymphoma requiring treatment, who have failed, unable to tolerate, or refused other available active therapies; patients should not have other treatment options considered curative (NOTE: for patients with lymphoma without CNS involvement, a re-biopsy is necessary unless the patient has had a previous biopsy =< 6 months prior to treatment on this protocol if there has been no intervening treatment; patients with biopsy-proven CNS lymphoma at any time are not required to have a rebiopsy to be eligible for this study); NOTE: relapsed NHL is defined as NHL that relapses after at least one prior therapy and does not have available curative therapy; refractory NHL is defined as NHL that has progressed or not responded to most recent therapy and has had at least one prior therapy and have no available curative therapies
* Measurable disease by CT or MRI or the CT portion of the PET/CT: must have at least one lesion that has a single diameter of >= 2 cm or tumor cells in the blood >= 5 x 10^9/L; skin lesions can be used if the area is >= 2 cm in at least one diameter and photographed with a ruler
* The following disease types are eligible: transformed lymphomas: diffuse large B cell lymphoma, mantle cell lymphoma, follicular lymphoma grade III; precursor B lymphoblastic leukemia/lymphoma; mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma/leukemia; precursor T-lymphoblastic leukemia/lymphoma; primary cutaneous anaplastic large cell lymphoma; anaplastic large cell lymphoma - primary systemic type; small lymphocytic lymphoma/chronic lymphocytic leukemia; follicular lymphoma, grades 1, 2; extranodal marginal zone B-cell lymphoma of MALT type; nodal marginal zone B-cell lymphoma; splenic marginal zone B-cell lymphoma; peripheral T cell lymphoma, unspecified; anaplastic large cell lymphoma (T and null cell type); lymphoplasmacytic lymphoma (Waldenstrom Macroglobulinemia); CNS lymphoma; post transplant lymphoproliferative disorders; mycosis fungoides/Sezary syndrome; primary effusion lymphoma; blastic NK-cell lymphoma; adult T-cell leukemia/lymphoma; extranodal NK/T-cell lymphoma, nasal type; enteropathy-type T-cell lymphoma; hepatosplenic T-cell lymphoma; subcutaneous panniculitis-like T-cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma - primary cutaneous type
* For lymphoplasmacytic lymphoma patients without measurable lymphadenopathy, measurable disease can be defined by both of the following criteria: bone marrow lymphoplasmacytosis with > 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy and quantitative IgM monoclonal protein > 1,000 mg/dL
* ANC >= 1000/uL
* Hgb >= 9 g/dl
* PLT >= 75,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN the direct bilirubin must be normal
* AST =< 3 x ULN
* Albumin > 3.0 g/dl
* Creatinine =< 2.5 x ULN
* Serum potassium, magnesium and phosphorus >= LLN and =< 1.2 x ULN
* Total serum calcium [corrected for serum albumin] or ionized calcium >= LLN
* Clinically euthyroid; patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
* Baseline MUGA or ECHO must demonstrate LVEF >= the lower limit of the institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to return to Mayo Clinic
* Life expectancy >= 12 weeks
* Willingness to provide blood and tissues samples for research studies as required by the protocol
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* ECOG performance status (PS) 0, 1 or 2

Exclusion Criteria

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Candidate for known standard therapy for the patient's disease that is potentially curative
* Uncontrolled infection requiring ongoing antibiotics
* Any prior therapy for lymphoma within the previous 2 weeks for standard treatments and within 4 weeks for experimental therapies unless the patient has recovered from the nadir of the previous treatment to a level that meets the inclusion criteria
* Receiving corticosteroids > 20mg of prednisone per day (or equivalent)
* Persistent toxicities >= grade 2 from prior chemotherapy or biological therapy regardless of interval since last treatment
* Patients with congenital long QT syndrome
* History or presence of sustained ventricular tachyarrhythmia (patients with a history of atrial arrhythmia are eligible but should be discussed with the study PI prior to enrollment)
* Any history of ventricular fibrillation or torsade de pointes
* Bradycardia defined as HR < 50 bpm; patients with pacemakers are eligible if HR >= 50 bpm
* Screening ECG with a QTcFredericia (QTcF) > 450 msec
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Patients with myocardial infarction or unstable angina =< 6 months prior registration
* Other clinically significant heart disease (e.g. CHF NY Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Pregnant women or women of reproductive ability who are unwilling to use effective contraception during the study and for 3 months after stopping treatment
* Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 3 months after stopping treatment
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation); patients should have recovered from any immunotherapy, chemotherapy, or radiation therapy related toxicities
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C with uncontrolled disease; baseline testing for HIV and hepatitis C is not required
* Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea > CTCAE Grade 2, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Any severe and/or uncontrolled medical conditions or other conditions that, in the treating physician's opinion, could adversely impact their ability to participate in the study; patients on chronic oxygen therapy, those with liver disease such as cirrhosis, chronic hepatitis or chronic persistent hepatitis, or uncontrolled infections will be excluded
* Concomitant use of strong or moderate CYP3A4 inhibitors
* Using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Active bleeding tendency. NOTE: Patients on therapeutic anticoagulation should be monitored carefully to maintain therapeutic level of anticoagulation to avoid increased risk of bleeding due to concurrent drug induced thrombocytopenia. It is suggested that patients who require anticoagulation therapy while on therapy use low molecular weight heparin (LMWH).
* Major surgery =< 4 weeks prior to registration or have not recovered from side effects of such therapy
* History of other prior malignancies except for properly treated basal cell or squamous cell carcinoma of skin, in situ cervical cancer, in situ breast cancer or early stage prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Johnston, M.D., Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (LBH589): Patients receive oral 40 mg panobinostat 3 times weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (LBH589)
Started | 41
Completed | 39
Not Completed | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are summarized for patients who completed the study.
Arm/Group | Arm I (LBH589)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 61.0 [37.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Responses Defined to be a CR or PR Noted as the Objective Status
Description: The primary endpoint of this phase II trial is the proportion of confirmed responses (complete response (CR) or partial response (PR)) noted as the objective status and will be considered synonymous with "success" for this study.Response will be evaluated using all cycles of treatment. A CR is defined using the Cheson et al. Revised Response Criteria for Malignant Lymphoma as Disappearance of all evidence of disease. A PR is defined as Regression of measurable disease and no new sites with ≥50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients.
Time Frame: Every 28 days for up to 2 years
Population: Patients who completed the study were evaluable for the primary outcome. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
Measure: Number (95% Confidence Interval); unit: proportion of CR or PR patients
Arm/Group | Arm I (LBH589)
Number analyzed (Participants) | 39
proportion of CR or PR patients | 0.21 [0.07 to 0.38]

2. Secondary Outcome: Median Overall Survival Time
Description: The median overall survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Every 6 months for up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (LBH589)
Number analyzed (Participants) | 39
months | 14.9 [8.8 to 46.4]

3. Secondary Outcome: Median Progression-free Survival Time
Description: The median progression-free survival time is defined as the time from registration to progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. Progression is defined using the Cheson et al. Revised Response Criteria for Malignant Lymphoma as: Any new lesion or increase by ≥50% of previously involved sites from nadir, Appearance of a new lesion(s) > 1.5 cm in any axis, ≥50% increase from nadir in SPD of more than one node, or ≥50% increase in longest diameter of a previously identified node > 1 cm in short axis, Lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy, > 50% increase from nadir in the SPD of any previous lesions, New or recurrent involvement.
Time Frame: Every 6 months for up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (LBH589)
Number analyzed (Participants) | 39
months | 3.1 [2.0 to 8.4]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression (PD) is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir).
Time Frame: Every 6 months for up to 2 years
Population: Patients who achieved a confirmed response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (LBH589)
Number analyzed (Participants) | 8
months | 19.7 [15.1 to 28.1]

5. Other Pre Specified Outcome: Pharmacokinetic/Pharmacodynamic of LBH589 and Correlation With Clinical Effects as Assessed by Immunoblotting, SNPs Analysis, Serum Cytokine Assays, and Flow Cytometry for Suppressive Monocytes (Correlative Studies)
Time Frame: At baseline and day 1 of courses 3, 5, 7 and every three courses thereafter for up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Arm I (LBH589)
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 34/41
Other Adverse Events (participants affected / at risk) | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (LBH589) (N=41)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 3 (7)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 12 (18)
Platelet count decreased (Investigations) | 33 (46)
Serum amylase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (LBH589) (N=41)
Anemia (Blood and lymphatic system disorders) | 11 (20)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 31 (98)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 29 (63)
Vomiting (Gastrointestinal disorders) | 15 (20)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 35 (159)
Lung infection (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (7)
Alkaline phosphatase increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 2 (2)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (7)
Lymphocyte count decreased (Investigations) | 6 (8)
Neutrophil count decreased (Investigations) | 17 (83)
Platelet count decreased (Investigations) | 19 (61)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 15 (47)
Anorexia (Metabolism and nutrition disorders) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (18)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 4 (15)
Headache (Nervous system disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (4)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes